CLINICAL TRIAL: NCT04430621
Title: Effects of Follicle-Stimulating Hormone Injection on Flow Mediated Dilation in Healthy Males
Brief Title: Effects of FSH on Endothelial Function (FEND)
Acronym: FEND
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, RAFFAELE NAPOLI, Associate Professor, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FSH1
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Change in Flow Mediated Dilation
Keywords: endothelial function, atherosclerosis, FSH, FMD
MeSH Terms: conditions — Atherosclerosis | interventions — Follicle Stimulating Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FSH (Experimental): FSH, 300 IU s.c.
  Interventions: Drug: Follicle Stimulating Hormone
- Control (Placebo Comparator): Placebo, s.c.
  Interventions: Drug: Follicle Stimulating Hormone

INTERVENTIONS:
Drug: Follicle Stimulating Hormone — FSH will be administered s.c. in the morning to male healthy subjects

SUMMARY:
Purpose of the study will be to evaluate the effects of the s.c. administration of 300 IU of FSH in 16 healthy males. The endothelial function will be evaluated by the measurement with ecographic approach of the flow mediated dilation (FMD) of the brachial artery. The FMD will be measured before and 6, 12, 24 or 48 hours after FSH or placebo adiministration in the same subjects studied 2 weeks apart. The results will help to clarify whether perturbation of FSH, similar to the one observed in women after the menopause, affect endothelial function.

DETAILED DESCRIPTION:
The effects of follicle-stimulating hormone (FSH) have been poorly studied. In women, FSH is involved in estrogen production, while in men regulates spermatogenesis. On the other hand, in women, menopause is associated with an increase in the risk of cardiovascular disease and the concentration of FSH rises. It is unclear whether such an increase has any effect on the development of atherosclerosis. Endothelial dysfunction represents an early trigger of atherosclerosis. Since estrogens can directly stimulate endothelial function and increase in response to FSH administration, males might represent a potential model to study the effcts of FSH independent from estrogens.Purpose of the study will be to evaluate the effects of the s.c. administration of 300 IU of FSH in 16 healthy males. The endothelial function will be evaluated by the measurement with ecographic approach of the flow mediated dilation (FMD) of the brachial artery. The FMD will be measured before and 6, 12, 24 or 48 hours after FSH or placebo adiministration in the same subjects studied 2 weeks apart. The results will help to clarify whether perturbation of FSH, similar to the one observed in women after the menopause, affects endothelial function.

ELIGIBILITY:
Inclusion Criteria: Healthy volunteers -

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-08-10 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in flow mediated dilation | before and 48 hours after FSH or placebo administration
  Evaluation of endothelial function of the brachial artery

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Napoli, MD, Principal Investigator — University Federico II
Locations (1):
- Internal Medicine and Diabetes Unit, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No